CLINICAL TRIAL: NCT06084910
Title: Self-Concept Reinforcement for Early School Readiness: Pilot Randomized Controlled Trial of a Clinic-Based Intervention for Young African American Children
Brief Title: Self-Concept Reinforcement for Early School Readiness
Acronym: SCR4ESR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ashaunta Anderson, Assistant Professor of Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHLA-23-00279; 1K23MD016944-01A1 (NIH)
Record Dates: First submitted 2023-09-08; First posted 2023-10-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Child Behavior; Child Behavior Problem; Child Behavior Disorders
Keywords: Child Behavior; Literacy; Early Childhood; Parenting; Self-Concept
MeSH Terms: conditions — Child Behavior; Child Behavior Disorders; Literacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Caregiver-child dyads that receive the Self-Concept Reinforcement for Early School Readiness (SCR4ESR) intervention
  Interventions: Behavioral: Self-Concept Reinforcement for Early School Readiness; Behavioral: Reach Out and Read
- Treatment-As-Usual Control Group (Active Comparator): Caregiver-child dyads that receive standard Reach Out and Read intervention without additional emphasis on self-concept
  Interventions: Behavioral: Reach Out and Read

INTERVENTIONS:
Behavioral: Self-Concept Reinforcement for Early School Readiness — Self-Concept Reinforcement for Early School Readiness (SCR4ESR) is based on the nationwide Reach Out and Read (ROR) program adapted to reinforce self-concept. ROR provides children's books, brief book-sharing advice, and developmental surveillance at pediatric well child visits. Each of the 5 SCR4ESR sessions provides 1 children's book with a self-concept theme, 1 parent handout, and modeling of book-sharing.
  Other Names: SCR4ESR
  Arms: Experimental Group
Behavioral: Reach Out and Read — ROR provides children's books and brief book-sharing advice at pediatric well child visits
  Other Names: ROR

SUMMARY:
The goal of this pilot randomized controlled trial is to evaluate a self-concept intervention (Self-Concept Reinforcement for Early School Readiness (SCR4ESR)) in young African American children using experimental and mixed methods. SCR4ESR provides self-concept themed children's books and advice at health supervision visits of children enrolled at ages 2-4 years.

The specific aims of the proposed project are to:

1. assess the feasibility and acceptability of SCR4ESR implementation among parents and providers,
2. evaluate the capacity of SCR4ESR to improve self-concept reinforcement and book-sharing behaviors in parents of young African American children, and 3) evaluate the capacity of SCR4ESR to improve behavioral health and literacy in young African American children. The interviews conducted in Aim 1 will guide refinement of the intervention tested in Aims 2 and 3.

The qualitative assessment will be complemented by quantitative trial statistics (e.g., recruitment rate) that inform trial feasibility and acceptability. Finally, the mechanism by which SCR4ESR impacts the primary outcome, behavioral health, and the secondary outcome, literacy, will be evaluated by structural equation modeling. This project will inform the development and implementation of early childhood interventions that improve the health of African Americans.

DETAILED DESCRIPTION:
Study Design. The proposed mixed methods study has 2 phases. Phase 1 will evaluate the feasibility and acceptability of SCR4ESR implementation from the perspectives of parents and providers (Aim 1, qualitative). Phase 2 will conduct a pilot randomized controlled trial (RCT) of SCR4ESR+ROR versus ROR alone in parents of 2- to 4-year-old African American children to assess SCR4ESR's impact on parenting behaviors, child behavioral health, and literacy; and to assess feasibility of the trial (Aims 2 & 3, quantitative).

Phase 1: Evaluation of the Feasibility and Acceptability of SCR4ESR (Aim 1).

Phase 1 will recruit 15 parents and 15 providers from 2 AltaMed clinics. Eligible parents will: 1) be 18 years old or older, 2) speak English, 3) be the legal guardian of a 2- to 4-year-old African American child, and 4) have experience with ROR. The exclusion criteria include parents whose target child has severe cognitive impairment or communication difficulties (i.e., severe intellectual disability or non-verbal). We will contact over 45 families over the 3-month recruitment period. The Principal Investigator (PI) will contact eligible parents 2 weeks prior to well child visits for recruitment purposes. Parents who provide informed consent by telephone will be scheduled for interviews following their children's well child visits. The informed consent form will be signed prior to interviews. The PI will also review next-day and day-of patient lists to identify potential participants. Study flyers will be posted at the clinic. The PI will recruit providers-including clinic leaders-through electronic mail and study flyers. Eligible providers must be board-certified pediatricians who completed an accredited residency program and have ROR experience. Sixty-minute key informant interviews will take place in a private space at the clinic. The PI will begin each 1-on-1 interview with a short instructional video on ROR. The PI will then give an overview of SCR4ESR, the self-concept book list, and parent handouts before asking prepared questions from the interview guide.Interview transcripts will be analyzed using standard qualitative methods.

Phase 2: Pilot Randomized Controlled Trial of SCR4ESR (Aims 2 and 3)

Aim 2: Test the capacity of SCR4ESR to improve proximal outcomes-self-concept reinforcement (SCR) and book-sharing behaviors-among parents of young African American children. Introduction. The objective of this aim is to examine the capacity of SCR4ESR to promote SCR and book-sharing behaviors in parents of 2- to 4-year-old African American children. We will test the working hypothesis that: 1) parents who receive SCR4ESR will exhibit more SCR and book-sharing behaviors than those who do not. Our approach to testing the working hypothesis will be to conduct a pilot RCT to determine the extent to which proximal intervention targets (SCR and book-sharing behaviors) are improved over a 15-month period of follow up within and between 2 groups (SCR4ESR+ROR and ROR alone). We will also quantitatively assess SCR4ESR feasibility and acceptability.

Aim 3: Test the capacity of SCR4ESR to improve exploratory distal outcomes-internalizing behaviors, externalizing behaviors, and literacy-in young African American children. Introduction. The objective of this aim is to examine the capacity of SCR4ESR to promote behavioral health and literacy in 2- to 4-year-old African American children. We will test the working hypotheses that: 1) children who receive SCR4ESR will exhibit better behavioral health and literacy than those who do not, and 2) the association between SCR4ESR and behavioral health and literacy will be mediated by parental SCR and book-sharing behaviors. Our approach to testing the working hypotheses will be to conduct a pilot RCT to determine the extent to which proximal intervention targets (SCR and book-sharing behaviors) act as mediators of improved distal targets (behavioral health and literacy) over a 15-month period of follow up within and between 2 groups (SCR4ESR+ROR and ROR).

Recruitment, Sampling Design, and Data Collection. Phase 2 will recruit caregivers of 134 children from 2 AltaMed clinics using the same methods we successfully employed during the preliminary study. Eligible parents will: 1) be 18 years old or older, 2) speak English, and 3) be legal guardian of the index 2- to 4-year-old African American child. The exclusion criteria include parents who: 1) have index children with severe cognitive impairment or communication difficulties (i.e., severe intellectual disability or nonverbal), 2) plan to move outside of the CHLA service area in the next 15 months, 3) are CHLA employees, or 4) participated in Aim 1 interviews. We expect to outreach to over 300 families during the 12-month recruitment period using a brief screening instrument. Potential parent-child dyads will be identified by the Research Coordinator (RC) who will review the list of patients scheduled for well child visits 2 weeks prior to each clinic day. Those who are unscheduled, but due for a well child visit will also be contacted. The remaining recruitment procedures are identical to those of Phase 1, including next-day and day-of screening, and appointment reminder phone calls.

Enrollment procedures. All consenting families will attend the enrollment well child visit with standard ROR. Then an RA (blinded to group assignment) will administer the baseline parent survey and child literacy assessment over 60 minutes. Next, a second RA will use the randomization module of the REDCap data capture system to randomize families in a 1:1 allocation to 1 of 2 trial arms stratified by clinic, age, and sex to: 1) SCR4ESR+ROR, or 2) ROR alone. If more than 1 child in a family meet inclusion criteria, 1 child will be randomly selected for participation. The blinded RA will remain responsible for subsequent assessments.

Experimental Group (SCR4ESR+ROR). Families assigned to the intervention will then receive SCR4ESR over 20 minutes (10 minutes content review, 10 minutes modeling book sharing, 1 children's book, and a parent handout) from the second RA (Table 5). SCR4ESR families will have a total of 5 intervention visits at 0, 3, 6, 9, and 12 months after enrollment focused on topics that support self-concept and shared book reading (Table 5) with repeat parent survey and child literacy assessment at 9 and 15 months after enrollment. The 15month survey will also assess intervention feasibility and acceptability items adapted from the qualitative items in Aim 1. Intervention visits are designed to overlap with well child visits where ROR is delivered. Due to the schedule of well child visits by age, children will receive different doses of ROR over the 15-month study period: 3 (24-, 30-, and 36- month visits) or 2 (30- and 36-, 36- and 48-, or 48- and 60-month visits) ROR doses.

Treatment-as-Usual Control Group: Families randomized to ROR alone (and those in SCR4ESR+ROR) will receive standard ROR book-sharing advice and 1 ROR children's book at 2 or 3 well child visits per the schedule of ROR doses discussed above. ROR books do not require specific images or narratives. Control families will complete the same parent surveys and child literacy assessments as intervention families at 0, 9, and 15 months after enrollment. Providers will not receive additional training in SCR4ESR or ROR to reduce the chance of contamination between study groups.

Analysis Plan. The Phase 2 analytic plan entails: 1) preliminary exploratory data analyses, 2) summaries of trial statistics, 3) analyses of SCR4ESR effects on proximal outcomes/mediators (SCR and book sharing) and distal outcomes (child behavioral health and literacy), 4) exploratory evaluations of mediation, and 5) exploratory evaluation of moderators (child sex, parenting stress, and parent ethnic identity). Preliminary exploratory data analyses will evaluate the distribution of each proximal outcome/mediator and distal outcome. If variables are not normally distributed, normalizing transformations will be attempted; rank-based non-parametric tests will be used if normalizing transformations are not successful. Evaluations of SCR4ESR intervention effects on proximal (Aim 2 SCR and book sharing) and distal (Aim 3 behavioral health and literacy) outcomes will involve group comparisons on follow-up assessments conducted by intent-to-treat (Table 6); participants will be evaluated within their randomized group, regardless of level of adherence. The randomized groups will be compared on the mean levels of outcomes assessed at 0-, 9- and 15-months post-randomization using mixed effects linear models. A group*time interaction will test if the intervention effects on changes in outcomes differ at 9 and 15 months. Significance testing will use a 2-sided P value of 0.05. Mediation analyses will use cross-lagged structural equation modeling (SEM) to evaluate: (1) the effect of SCR4ESR on the potential mediating variables (CPR measured in Hughes' Racial Socialization Scale and book-sharing behaviors measured in the book-sharing scale, (2) the associations of CPR and book sharing with subsequent distal outcomes (behavioral health and literacy), (3) the cross-lagged associations of behavioral health and literacy outcomes on subsequent CPR and book sharing, and (4) estimates of the direct effects (not through mediators) and indirect (mediated) effects of CPR4ESR on distal outcomes. Bias-corrected bootstrapped estimates and 95% CIs on the indirect (mediated) effects will be made. Covariates will include randomization stratification variables, age, gender, and clinic. Analyses will test for moderated mediation by gender.

Secondary Exploratory Moderator Analyses. All analyses will be stratified by potential moderators (child sex, parenting stress, and parent ethnic identity) separately. In the entire sample, interaction terms of group by moderator will test for differences in intervention effects among these subgroups. Although we will not have statistical power to test for moderator-intervention interactions, we will nonetheless conduct stratified analyses to identify moderator-specific SCR4ESR effects.

Statistical Power. Given pilot 25% attrition rate, we will recruit 134 participants to yield 100 to study end. For 100 participants, proportions will be estimated with a 95% CI width of 0.13-0.20 (again depending on the actual proportion estimate). For the sample size of 100 (50 per group), we computed the precision of the 95% CI for estimating 1-group means (e.g., for within-group mean change) and 2-group mean differences (for intervention effect sizes) on trial outcomes. We will be able to estimate 1-group mean changes with a 95% CI that is ±0.28SD (standard deviation), and 2-group mean differences with a 95% CI that is ±0.40SD. This pilot trial is not designed to statistically detect intervention group differences on outcomes. Nonetheless, the sample size of 50 per group will allow detection of group differences with medium Cohen's d effect sizes (mean group difference/SD) of 0.57 and higher (at 80% power, 2-sided alpha=0.05) and withingroup Cohen's d effect sizes of 0.40 and higher. The sample size of 100 will also allow for detection of correlations (e.g., between proximal and distal outcomes) of 0.28 and higher at 80% power.

Expected Outcomes. We expect the mixed methods study of SCR4ESR feasibility and acceptability will allow us to improve the intervention and trial. We will gain exploratory insight into the mechanism relating SCR4ESR to behavioral health and literacy in young African American children and present findings to the CAB in Year 4.

Potential Problems and Alternative Strategies.Recruitment is a potential problem that will be addressed with a 12-month recruitment period, proactive searches for potential participants, and incentives (i.e., $20 Amazon gift cards at first 3 visits, $40 gift cards at next 3 visits, and $20 transportation stipend for each visit). Sample size may also be limited by dropout.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Legal guardian must be 18 years old or older
* Speak English
* Legal guardian of the index 2 to 4-year-old African American child

Exclusion Criteria:

* Index child has severe cognitive impairment or communication difficulties (i.e., severe intellectual disability or nonverbal)
* Plan to move outside of the Children's Hospital Los Angeles (CHLA) service area in the next 15 months
* CHLA employee
* Participated in Aim 1 interviews

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline for externalizing behavior score for Child Behavioral Health as measured by Child Behavior Checklist | Baseline to 15 months post-enrollment
  Child Behavior Checklist - Externalizing behaviors. Items rated on a Likert scale from 0 to 2. The items are divided across categories and summed by category such that higher sums amount to more behavioral problems. 2-3 years old: minimum/maximum scores 0 to 128. 4 years and older: minimum/maximum scores 0 to 236.
Mean change from baseline for internalizing behavior score for Child Behavioral Health as measured by Child Behavior Checklist | Baseline to 15 months post-enrollment
  Child Behavior Checklist - internalizing behaviors. Items rated on a Likert scale from 0 to 2. The items are divided across categories and summed by category such that higher sums amount to more behavioral problems. 2-3 years old: minimum/maximum scores 0 to 128. 4 years and older: minimum/maximum scores 0 to 236.

SECONDARY OUTCOMES:
Mean change from baseline for Child Early Language Skills using the Receptive One-Word Picture Vocabulary Test. | Baseline to 15 months post-enrollment
  Receptive One-Word Picture Vocabulary Test (ROWPVT.) Respondents select 1 picture among 4 that best represents the word spoken by the examiner; this repeats until a set number of consecutive errors. Therefore, higher score suggests better literacy.
Mean change from baseline for Child Early Literacy Skills using the The Reading House for participants 3-5 years old. | Baseline to 15 months post-enrollment
  The Reading House uses a children's book to screen for emergent literacy skills. The assessor shares the book with the child and screens skills using a 9-item, scripted scoring form.
Mean change from baseline for Bookreading Quantity Subdimension using STIMQ 2-READ Scale | Baseline to 15 months post-enrollment
  STIMQ 2-READ Scale. Book-sharing scale (scale to assess ways caregiver shares books with child). 12-35 months old: minimum/maximum scores are 0 to 9. 36 months and older: minimum/maximum scores are 0 to 9. Higher scores indicate more book-reading behaviors.
Mean change from baseline for Diversity of Content/Concepts using STIMQ 2-READ Scale. | Baseline to 15 months post-enrollment
  STIMQ 2-READ Scale. Book-sharing scale (scale to assess ways caregiver shares books with child). 12-35 months old: minimum/maximum scores are 0 to 6. 36 months and older: minimum/maximum scores are 0 to 8. Higher scores indicate more book-reading behaviors.
Mean change from baseline Bookreading Quality Subdimension using STIMQ 2-READ Scale. | Baseline to 15 months post-enrollment
  STIMQ 2-READ Scale. Book-sharing scale (scale to assess ways caregiver shares books with child). 12-35 months old: minimum/maximum scores are 0 to 4. 36 months and older: minimum/maximum scores are 0 to 5. Higher scores indicate more book-reading behaviors.
Mean change from baseline Self-Concept Reinforcement using Hughes' Socialization Scale. | Baseline to 15 months post-enrollment
  Hughes' Socialization Scale. Three items rated on Likert scale from 0 to 5 and summed such that higher score suggests more self-concept reinforcement. Minimum to maximum summed scores are 0 to 15.

OTHER OUTCOMES:
Book-sharing beliefs | 0 and 15 months
  Parental Reading Belief Inventory (PRBI)

CONTACTS AND LOCATIONS:
Overall Officials: Ashaunta T Anderson, MD, MPH, MSHS, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
I am working on delineating the plan that would facilitate IPD sharing. Adequate resources need to be allocated to make it possible.

REFERENCES:
- [Background] Anderson AT, Luartz L, Heard-Garris N, Widaman K, Chung PJ. The Detrimental Influence of Racial Discrimination on Child Health in the United States. J Natl Med Assoc. 2020 Aug;112(4):411-422. doi: 10.1016/j.jnma.2020.04.012. Epub 2020 Jun 10. PMID 32532525
- [Background] Lee RT, Perez AD, Boykin CM, Mendoza-Denton R. On the prevalence of racial discrimination in the United States. PLoS One. 2019 Jan 10;14(1):e0210698. doi: 10.1371/journal.pone.0210698. eCollection 2019. PMID 30629706
- [Background] Priest N, Paradies Y, Trenerry B, Truong M, Karlsen S, Kelly Y. A systematic review of studies examining the relationship between reported racism and health and wellbeing for children and young people. Soc Sci Med. 2013 Oct;95:115-27. doi: 10.1016/j.socscimed.2012.11.031. Epub 2012 Dec 19. PMID 23312306
- [Background] Breslau J, Kendler KS, Su M, Gaxiola-Aguilar S, Kessler RC. Lifetime risk and persistence of psychiatric disorders across ethnic groups in the United States. Psychol Med. 2005 Mar;35(3):317-27. doi: 10.1017/s0033291704003514. PMID 15841868
- [Background] Breslau J, Aguilar-Gaxiola S, Kendler KS, Su M, Williams D, Kessler RC. Specifying race-ethnic differences in risk for psychiatric disorder in a USA national sample. Psychol Med. 2006 Jan;36(1):57-68. doi: 10.1017/S0033291705006161. Epub 2005 Oct 5. PMID 16202191
- [Background] Campbell SB, Shaw DS, Gilliom M. Early externalizing behavior problems: toddlers and preschoolers at risk for later maladjustment. Dev Psychopathol. 2000 Summer;12(3):467-88. doi: 10.1017/s0954579400003114. PMID 11014748
- [Background] Stevenson J, Richman N, Graham P. Behaviour problems and language abilities at three years and behavioural deviance at eight years. J Child Psychol Psychiatry. 1985 Mar;26(2):215-30. doi: 10.1111/j.1469-7610.1985.tb02261.x. PMID 3980611
- [Background] Brooks-Gunn J, Markman LB. The contribution of parenting to ethnic and racial gaps in school readiness. Future Child. 2005 Spring;15(1):139-68. doi: 10.1353/foc.2005.0001. PMID 16130545
- [Background] Bannon WM, McKay MM, Chacko A, Rodriguez JA, Cavaleri M. Cultural Pride Reinforcement as a Dimension of Racial Socialization Protective of Urban African American Child Anxiety. Fam Soc. 2009;90(1):79-86. doi: 10.1606/1044-3894.3848. PMID 20046919
- [Background] McHale SM, Crouter AC, Kim JY, Burton LM, Davis KD, Dotterer AM, Swanson DP. Mothers' and fathers' racial socialization in African American families: implications for youth. Child Dev. 2006 Sep-Oct;77(5):1387-402. doi: 10.1111/j.1467-8624.2006.00942.x. PMID 16999806
- [Background] Caughy MO, Owen MT. Cultural socialization and school readiness of African American and Latino preschoolers. Cultur Divers Ethnic Minor Psychol. 2015 Jul;21(3):391-9. doi: 10.1037/a0037928. Epub 2014 Nov 3. PMID 25364832
- [Background] Caughy MO, O'Campo PJ, Randolph SM, Nickerson K. The influence of racial socialization practices on the cognitive and behavioral competence of African American preschoolers. Child Dev. 2002 Sep-Oct;73(5):1611-25. doi: 10.1111/1467-8624.00493. PMID 12361322
- [Background] Woods-Jaeger B, Briggs EC, Gaylord-Harden N, Cho B, Lemon E. Translating cultural assets research into action to mitigate adverse childhood experience-related health disparities among African American youth. Am Psychol. 2021 Feb-Mar;76(2):326-336. doi: 10.1037/amp0000779. PMID 33734798
- [Background] Anderson AT, Jackson A, Jones L, Kennedy DP, Wells K, Chung PJ. Minority Parents' Perspectives on Racial Socialization and School Readiness in the Early Childhood Period. Acad Pediatr. 2015 Jul-Aug;15(4):405-11. doi: 10.1016/j.acap.2014.11.002. Epub 2014 Dec 19. PMID 25534762
- [Background] Jones VF, Franco SM, Metcalf SC, Popp R, Staggs S, Thomas AE. The value of book distribution in a clinic-based literacy intervention program. Clin Pediatr (Phila). 2000 Sep;39(9):535-41. doi: 10.1177/000992280003900905. PMID 11005367
- [Background] Mendelsohn AL, Cates CB, Weisleder A, Berkule Johnson S, Seery AM, Canfield CF, Huberman HS, Dreyer BP. Reading Aloud, Play, and Social-Emotional Development. Pediatrics. 2018 May;141(5):e20173393. doi: 10.1542/peds.2017-3393. Epub 2018 Apr 9. PMID 29632254
- [Background] Garner A, Yogman M; COMMITTEE ON PSYCHOSOCIAL ASPECTS OF CHILD AND FAMILY HEALTH, SECTION ON DEVELOPMENTAL AND BEHAVIORAL PEDIATRICS, COUNCIL ON EARLY CHILDHOOD. Preventing Childhood Toxic Stress: Partnering With Families and Communities to Promote Relational Health. Pediatrics. 2021 Aug;148(2):e2021052582. doi: 10.1542/peds.2021-052582. PMID 34312296
- [Background] Shaw DS, Mendelsohn AL, Morris PA. Reducing Poverty-Related Disparities in Child Development and School Readiness: The Smart Beginnings Tiered Prevention Strategy that Combines Pediatric Primary Care with Home Visiting. Clin Child Fam Psychol Rev. 2021 Dec;24(4):669-683. doi: 10.1007/s10567-021-00366-0. Epub 2021 Sep 9. PMID 34505232
- [Background] Garcia Coll C, Lamberty G, Jenkins R, McAdoo HP, Crnic K, Wasik BH, Vazquez Garcia H. An integrative model for the study of developmental competencies in minority children. Child Dev. 1996 Oct;67(5):1891-914. PMID 9022222